CLINICAL TRIAL: NCT02477722
Title: Neurofeedback Preventive Intervention for PTSD: a Method to Strengthen Mental and Emotional Resilience
Brief Title: Neurofeedback Prevention For Early Stress Related Adversity
Acronym: NFPES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0616-14-TLV
Record Dates: First submitted 2015-05-31; First posted 2015-06-23 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Feedback, Psychological; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFP-NF (Experimental): Subjects are asked to change their brain activity in response to feedback they receive from the brain itself, mediated via various visual or auditory stimuli.
  Interventions: Other: EFP-NF
- Sham-NF (Sham Comparator): Placebo
  Interventions: Other: Sham

INTERVENTIONS:
Other: EFP-NF
  Arms: EFP-NF
Other: Sham
  Arms: Sham-NF

SUMMARY:
Exposure to life threatening, traumatic and stress inducing events in general is an inevitable part of military combat service . Among individuals exposed to a traumatic event, approximately 85-90 % will develop a stress response from which they will recover without need for any medical intervention whatsoever. However, roughly 10-15 % will continue to suffer from post-traumatic symptoms along with depression or anxiety disorders1, . The prominent symptoms of post - traumatic stress disorder (PTSD), consists of reliving the event via invasive and painful memories that include: images, thoughts or feelings, night terrors, and extreme emotional distress that arise when exposure to external or internal cues similar to or symbolizing aspects of the traumatic event. Following this distress, behavioral avoidance of situations that trigger unpleasant memories may develop. Such mental stress may lead to avoidance of social situations and hinder normal daily functioning in a variety of contexts2. The question arises as to what distinguishes between those who are exposed to a traumatic event and recover spontaneously and those who fail to resume daily life and develop PTSD. Attempts to find personality and environmental risk factors for the development of PTSD have yet to yield any unequivocal conclusions. This has lead the scientific community to look for neuro-physical risk factors as well . Furthermore, evidence that early diagnosis and treatment of the disorder helps reduce the severity of post-trauma symptoms -stresses the need for the accurate localization of neurological risk factors and new immediate and/or preventative interventions. The aim of the present project is to develop a brain oriented training method for early preventive interventions of PTSD.

DETAILED DESCRIPTION:
The most significant disadvantage of the current EEG-NF method is the low spatial resolution of the EEG, which does not allow for the localization of site activity within deep brain regions known to be associated with the development of PTSD, such as the amygdala, the hippocampus, and the mPFC. The aim of the present project is to overcome this drawback by integrating EEG and fMRI imaging methods, such that the patient will receive real-time feedback regarding the activation of emotional target areas located deep within the brain. FMRI is based on the measurement of metabolic changes following electrical activity in the brain, thus non-invasively representing the neuronal activity of various brain regions when performing emotional and/or cognitive tasks. fMRI has high spatial resolution, and in contrast to EEG - it allows for the localization of regions deep within the brain, such as those related to trauma responses within the limbic system and prefrontal cortex. Recently, real-time fMRI (rt fMRI) has been used to train subjects to modulate activity within deep brain regions , . Some studies have even shown that subjects can be trained to regulate activity within a network of regions including the mPFC and limbic regions, resulting in a positive effect on patients suffering from chronic pain and depression . Moreover, it has also been found that via real-time fMRI feedback subjects can be trained to regulate activity within networks that have been linked to emotional regulation; a skill critical for dealing with traumatic events . The major disadvantage of this method is that fMRI tests are expensive and inconvenient for the patient, and the MRI machine required for this method are stationary and not easily accessible.

To combine the advantages of both methods the investigators performed simultaneous testing of both EEG and fMRI. Using special algorithms, with high reliability, the investigators studied the electrical signals that represent activity related to emotional regulation within deep brain regions . This combination allowed for a significant improvement in the spatial resolution of the EEG device and added significant temporal information taken from the fMRI signal. The combined recording of EEG and fMRI with advanced computational methods, such as cross correlation and machine learning, provide significant improvement in the attribution of EEG signal localization, which until now could not be achieved with adequate reliability. In other words, the EEG pattern of activity reliably represents activation of deep limbic regions providing an "electrical fingerprint" (EFP) of these areas.

Accordingly, the investigators developed an innovative treatment protocol in which subjects are asked to control either visual or auditory stimuli, determined by feedback from the brain, based on the extent of the EFP . In a pilot study on a group of civilians the investigators showed that subjects successfully learned to modify their electrical brain signal based on the EFP . In an additional study, simultaneous recordings of EEG and fMRI showed that success was indeed related to changes in activity within deep brain regions involved in emotional regulation; such as the mPFC and hippocampus. Furthermore, our results indicate that following training to volitionally regulate the EFP via EEG-NF, participants exhibited improved emotion regulation .

Rationale for current study:

Based on the EFP model and the NF literature in the treatment of PTSD this study aims to examine the efficiency of an fMRI-guided-EEG-protocol for self-regulation through NF for reducing stress vulnerability.

The study will assign two groups:

experimental group: EFP neurofeedback control groups: Sham neurofeedback In order to assess the efficiency of the NF protocol as a preventative intervention for PTSD, the investigators plan to compare this treatment outcomes to those of a placebo sham protocol.

Primary objective:

Examine the efficiency of NF in reducing stress vulnerability.

Secondary objective:

Examine the efficiency of amygdala targeted Neurofeedback (NF) in reducing stress symptoms among individuals who were recently exposed to a traumatic event. .

Study design:

Randomized parallel design, with 2 groups: EFP-NF (n=35), Sham-NF (n=35)

Participant selection:

The study will involve 40 participants with PTSD symptoms between the ages of 18-40, who will be divided randomly into 2 groups (experimental group, control group).

Number of participants:

The study will involve 70 individuals.

Recruitment process:

Participants will be recruited from the ER and trauma clinic at TASMC. The hospital will provide our research team with daily lists of the individuals who arrived at the ER over the past 24 hours, screened for possible trauma related incidents. Our team will then contact the potential subjects over the phone and will request informed consent to conduct a phone interview to assess the presence of acute stress symptoms. A brief description of the study will be provided. If the individual agrees and is found suitable for further participation they will be invited to the trauma clinic at TASMC where a trained clinical psychologist will conduct a comprehensive PTSD evaluation. The trauma clinic at TASMC will also refer suitable patients from within their database for participation in our study. All subjects referred by the trauma clinic will undergo identical procedures for obtaining informed consent and subsequent clinical evaluation as those described above.

Intervention arms:

The study will include 2 groups. The experimental group will receive EEG-NF sessions targeted on the amygdalae and the control group will Sham-NF.

Brain area/s of interest:

The regions of interest will include the limbic system and more specifically the Amygdala, hippocampus ventral striatum, as well as cortical areas associated with emotional regulation (such as dorso-lateral PFC and dorso and ventro-medial PFC cingulated cortex and insula).

Study procedures:

Pre treatment phase Day 1 Participants will undergo a psychiatric evaluation (using SCID), and medication monitoring. Participants will also be asked to fill in demographic and psychological questionnaires assessing emotion regulation abilities (ERQ), state anxiety and traits (STAI), and questionnaires measuring symptoms of stress, anxiety and depression (CAPS, PCL, BDI).

Day 2 All Participants will undergo a brain-imaging scan to characterize brain network responses associated with emotional arousal and regulation. Participants will be scanned for functional and structural MRI which will include ROI localizer for the NF, resting state, emotional conflict task, facial recognition task reward task and DTI.

The research staff will explain the course of the MRI testing to the participant, and will enter with the subject into the mock simulator to verify that he is lying on his back properly and feels comfortable. During testing the patient will be presented with visual and auditory stimuli, as well as short video clips. Auditory presentation: stimuli will be heard via MRI-compatible headphones. Visual displays: the subject will view the stimuli through a mirror and projected onto a screen in the magnet room. In between sessions the patient will be given time to rest. Participants will be asked to avoid moving as much as possible during the scans.

The total duration of testing, from subject arrival to departure, will take approximately 90-180 minutes (20-30 minutes to fill out forms and undergo training, 30 minutes for explanations and a break, and 60 minutes of imaging). Participants will remain in the MRI for about 60 minutes, and under no circumstances will remain longer than 90 minutes.

Training phase The duration of the training phase will be 4 weeks. At this point participants will be randomly assigned to either the EFP-NF or T/A-NF groups. Both the EFP-NF and the T/A-NF groups will receive 1-2 sessions per week for a total of 6 sessions.

During training sessions, participants will train to develop skills for regulating brain activity using auditory or visual feedback. Each session will last an hour, including EEG Cap placement and filling state questionnaires. The participant will be seated comfortably in front of a computer screen. A staff member will explain the goal of the meeting to the participant, introduce the equipment to be used, and describe the course of the meeting. Following the above explanations, the staff member will place the EEG cap on the participant's head and will ensure that the participant feels comfortable. The EEG - Neurofeedback practice will consist of five-minute segments repeated for up to 30 minutes. During each practice segment the participant will be asked to modify any visual or auditory media that provides feedback on the degree of successful brain training. For example, during visual feedback the participants will be asked to lower the speed of a skateboard presented on the computer screen or alternatively, during auditory feedback to reduce the level of music audible through headphones placed on their ears. After every two practice segments, the duration of each practice will increase such that the two first steps will be very short (about 5 minutes each) and the last two the longest (about 10 minutes each); a total of six steps every trial over a total of approximately 45 minutes

Post treatment phase This phase will take place 3-5 days after the end of the training phase. Day 1

* Participants will undergo a second psychological evaluation (CAPS).
* Participants will complete the same questionnaires as in the pre treatment phase (BDI, ERQ, STAI, PCL).

Day 2 • All Participants will be scanned for functional and structural MRI which will include ROI localizer, resting state, DTI.

Follow-up phase Day 1-5

• All participants will receive 2 maintenance sessions (EFP-NF or T/A-NF)

Day 6

* Participants will undergo a third psychological evaluation (CAPS).
* Participants will complete the same questionnaires as in the previous phases (BDI, ERQ, STAI, PCL).

Data collection:

Researchers will assist participants filling in the electronic questionnaires and will conduct the non electronic ones (these would be later transcribed to excel sheets by research assistants).

Researchers will run the MRI scans and the NF sessions (all the rt-fMRI NF and some of the EFP-NF), together with two to five research assistants. The contact with the participants will be by E-mail and phone. The research assistants will monitor participation. The participants will receive a reminder (by phone and or email) one day prior to each session.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to traumatic event in the past 14 days. Standard criteria for inclusion in medical MRI scans, according to the procedures set forth at MRI Medical Center in Tel - Aviv Sourasky will be applied to all participants.

Exclusion Criteria:

* Standard criteria for exclusion in medical MRI scans, according to the procedures set forth at MRI Medical Center in Tel - Aviv Sourasky will be applied to all participants and in accordance with the "metal form". For example, metal that cannot be removed, Orthodontal accessories connected to ones teeth, or current systemic diseases (including chronic diseases).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in Psychiatric Evaluation of PTSD Symptoms | Days 1-7 and 6 months after training

SECONDARY OUTCOMES:
fMRI Scan as a measure of change in amygdala reactivity | Days 1-7 and 6 months after training
Change in Emotion Regulation Questionnaire (ERQ) as a measure of change in cognitive coping strategies | Days 1-7 and 6 months after training
State/Trait Anxiety Inventory (STAI) as a measure of change in state & trait anxiety | Days 1-7 and 6 months after training
Beck Depression Inventory (BDI-II) as a measure of change in clinical depression | Days 1-7 and 6 months after training
Debriefing interview questionnaire as a measure of general experience of the process and adverse effects | 6 months after training
PCL as a measure of change in PTSD symptoms | Days 1-7 and 6 months after training
Emotional conflict task as a measure of change in facial recognition measuring emotional regulation | Days 1-7 and 6 months after training

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, M.D, Ph.D, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Whol Institute for Advanced Imaging, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Caria A, Veit R, Sitaram R, Lotze M, Weiskopf N, Grodd W, Birbaumer N. Regulation of anterior insular cortex activity using real-time fMRI. Neuroimage. 2007 Apr 15;35(3):1238-46. doi: 10.1016/j.neuroimage.2007.01.018. Epub 2007 Jan 31. PMID 17336094
- [Background] deCharms RC, Christoff K, Glover GH, Pauly JM, Whitfield S, Gabrieli JD. Learned regulation of spatially localized brain activation using real-time fMRI. Neuroimage. 2004 Jan;21(1):436-43. doi: 10.1016/j.neuroimage.2003.08.041. PMID 14741680
- [Background] deCharms RC, Maeda F, Glover GH, Ludlow D, Pauly JM, Soneji D, Gabrieli JD, Mackey SC. Control over brain activation and pain learned by using real-time functional MRI. Proc Natl Acad Sci U S A. 2005 Dec 20;102(51):18626-31. doi: 10.1073/pnas.0505210102. Epub 2005 Dec 13. PMID 16352728
- [Background] Linden, D. & Lancaster, T. (2011). Functional magnetic resonance imaging (fMRI) - based neurofeedback as a new treatment tool for depression. European Psychiatry, 26(1), 937-946.
- [Background] Johnston SJ, Boehm SG, Healy D, Goebel R, Linden DE. Neurofeedback: A promising tool for the self-regulation of emotion networks. Neuroimage. 2010 Jan 1;49(1):1066-72. doi: 10.1016/j.neuroimage.2009.07.056. Epub 2009 Jul 29. PMID 19646532
- [Background] Meir-Hasson Y, Kinreich S, Podlipsky I, Hendler T, Intrator N. An EEG Finger-Print of fMRI deep regional activation. Neuroimage. 2014 Nov 15;102 Pt 1:128-41. doi: 10.1016/j.neuroimage.2013.11.004. Epub 2013 Nov 15. PMID 24246494
- [Background] Cavazza, M. et al., Towards emotional regulation through neurofeedback, in Proceedings of the 5th Augmented Human International Conference (ACM, March, 2014), p. 42.
- [Background] Meir-Hasson, Y. et al., A Common amygdala EEG Finger-Print for self-regulation training, (Submitted). Journal of Neuroscience Methods.
- [Background] Keynan, J.N., et al.,. Reaching the unreachable: online-monitoring and guided regulation of amygdala activity using spatially enriched EEG. (In Preparation).